CLINICAL TRIAL: NCT04437277
Title: Screening for Chronic Hepatitis C Virus in Hospitalized Patients at Saint Joseph Hospital in Marseille
Brief Title: Screening for Chronic Hepatitis C Virus in Hospitalized Patients
Acronym: DeViCHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-A02595-50
Record Dates: First submitted 2020-01-06; First posted 2020-06-18 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Monocentric interventional longitudinal risk and minimal constraint study, consenting and consecutive in-patients recruited within the hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients consenting (Experimental)
  Interventions: Diagnostic Test: Hepatitis C, serology

INTERVENTIONS:
Diagnostic Test: Hepatitis C, serology — Inclusion of patients in conventional hospitalization at Saint Joseph Hospital. Each consenting patient benefits from a screening HCV serology carried out during a biological sample indicated by his state of health. In the case of positive HCV serology, an additional sample will be taken in search of viral replication. All detectable HCV PCR patients will be admitted to hepatology consultation for assessment of liver status including non-invasive methods and possible treatment according to the conditions of the Marketing Authorization and recommendations for routine clinical practice. Data on management (treatment or non-treatment and treatment outcome: prolonged virological response 12 weeks after completion of treatment) will be collected.
  Other Names: Hepatitis C, PCR

SUMMARY:
Chronic viral hepatitis C is a public health problem and several management recommendations are available. According to the HAS, hepatitis C screening consists of a targeted screening of people at risk of infection by the virus, in particular to drug users, to people from countries with a high prevalence of the virus or who have received care in those countries, people transfused before 1992, or people who have been or have been imprisoned. Our study proposes to evaluate hepatitis C screening in consenting patients hospitalized in Saint Joseph. These previously identified patients with comorbidities will be cared for according to current national practices that reduce HCV morbidity and mortality.

DETAILED DESCRIPTION:
Hepatitis C screening is based on a blood test, in particular the Elisa test, which looks for anti-HCV antibodies. In the case of positive C viral serology, the search for the C virus from a blood test makes it possible to detect the genome (RNA) of the virus, which is thus directly detected by a so-called "PCR" technique. Although screening activity is important in France, it remains insufficient. In December 2016, HAS concluded that risk-based targeted screening has limitations and contributes to the persistence of a hidden epidemic of viral C infection. It is estimated that 75,000 people are unaware of being carriers of the hepatitis C virus. However, there is safe, effective and well-tolerated treatment. With duration of 8 to 12 weeks it allows a healing of HCV in more than 95% of subjects. AFEF recommendations aim to achieve viral elimination C (as early as 2025). This elimination is defined as a 90% decrease in new infections associated with a 65% reduction in HCV mortality. OMS has planned this target for 2030. To achieve this goal, a number of measures are gradually being implemented focusing on universal treatment and universal screening. The hospital may be a place where systematic screening is interesting. In 2017, the prevalence of anti-HCV positive antibodies in the facility, apart from the Hepato-Gastroenterology service, was 1.7%, more than twice the estimated prevalence in our general population. These data give a rationale for the realization of this study.

ELIGIBILITY:
Inclusion Criteria:

* all in-patient patients and consenting to participate at the study.

Exclusion Criteria:

* Refusal to participate in the study
* Contraindication to a blood sample (Impossibility of a peripheral venous approach and any clinical condition that may indicate a venous sample)
* Minor patient
* Patient unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of hepatitis C through the different department of Saint Joseph Hospital | one day
  At every hospitalized patients the trial will be presented. the viral screening will be proposed for the purpose of treating patients who will be viremic

SECONDARY OUTCOMES:
number of viremic patients with risk factors | one day
  Identify viremic patients enrolled with identified risk factors
number of viremic patients without risk factors | one day
  Identify viremic patients enrolled without identified risk factors
number of patients who refuse viral screening | one day
  study will be presented to all hospitalized patients in Saint Joseph Hospital but investigators will estimate pateints who refuse to participate

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Joseph, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No